CLINICAL TRIAL: NCT05479825
Title: Tubeless Intersegmentectomy Plane Identification With Inflation- Deflation Line Combined With Fluorography
Brief Title: Tubeless Intersegmentectomy Plane Identification With Fluorography
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Tubeless Intersegmental ICG
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-05

CONDITIONS: Operation Time; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- inflation- deflation line combined with ICG fluorography (Experimental): Identification of the intersegmental plane using inflation- deflation line combined with ICG fluorography under the status of tubeless
  Interventions: Procedure: inflation- deflation line combined with ICG fluorography

INTERVENTIONS:
Procedure: inflation- deflation line combined with ICG fluorography — Identification of the intersegmental plane using inflation- deflation line combined with ICG fluorography under the status of tubeless

SUMMARY:
Background: We aimed to evaluate the combination of inflation- deflation method and fluorography with the ICG injection in the tubeless minimally invasive segmentectomy (no intubation, VATS or Robotic).

Methods: A one- armed, prospective randomized controlled study was designed. The intersegmental plane was not so clear during the tubeless minimally invasive segmentectomy, and the presentation of the plane sometimes cost more time. This study will evaluate consecutive patients with the combination of inflation- deflation method and fluorography with the ICG injection.

ELIGIBILITY:
Inclusion Criteria:

1. cardio- pulmonary function can tolerate the minimally invasive surgery (including VATS and robotic surgery);
2. benign pulmonary lesion considering for segmentectomy;
3. ≤2cm pulmonary adenocarcinoma with ground- glass components, considering for segmentectomy.

Exclusion Criteria:

1. cardio- pulmonary function can not tolerate the minimally invasive surgery (including VATS and robotic surgery);
2. segmentectomy is not considered as the surgery plan.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
time of description and management of the intersegmental plane | during surgery
  time of description and management of the intersegmental plane
perioperative complication rate | within 7 days after surgery
  perioperative complication rate
incisal margin of the tumor | during surgery
  incisal margin of the tumor

SECONDARY OUTCOMES:
disease- free survival | within 5 years after surgery
  DFS

CONTACTS AND LOCATIONS:
Overall Officials: Xiaogang Zhao, doctor, Study Director — The Second Hospital of Shandong University
Locations (1):
- Yunpeng Zhao, Jinan, Other (Non U.s.), China